CLINICAL TRIAL: NCT04774575
Title: Randomized Controlled Multicentre Trial to Quantify the Benefits of Biomarkers in Routine Patient Care in Kidney Transplant Recipients" EU-TRAIN IMPACT Trial
Brief Title: Quantify the Benefits of Biomarkers in Routine Patient Care in Kidney Transplant Recipients
Acronym: EUTRAIN IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200984
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Renal Transplantation
Keywords: renal transplantation; non-invasive biomarkers; risk evaluation; randomized trial

STUDY DESIGN:
Intervention Model Description: This is a 12-month follow-up multicenter, randomized, biomarker strategy design trial, whereby kidney transplant patients will be randomized 1:1 at the time of transplantation in 2 study groups:
  * Group I ("routine group"): Patients will follow a standard clinical follow-up based on kidney allograft function (serum creatinine, estimated glomerular filtration rate (eGFR), proteinuria) and a surveillance allograft biopsies performed at 3 and 12 months after transplantation (M3 and M12).
  * Group II ("biomarker guided follow-up"): Patients will follow a biomarker-guided strategy based on specific non-invasive biomarkers as defined in EUTRAIN-1 study on the basis of its detection and prediction capacities for rejection at M3 to decide whether a biopsy is performed. At M12 a routine biopsy is performed.
  In both groups, a biopsy can be performed up on clinical decision if needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine group (No Intervention): Patients will follow a standard clinical follow-up based on kidney allograft function (serum creatinine, estimated glomerular filtration rate (eGFR), proteinuria) and a surveillance allograft biopsies performed at 3 and 12 months after transplantation (M3 and M12). Visits with biopsies for clinical indication are left to the appreciation of the investigator
- biomarker guided follow-up (Experimental): Patients will follow a biomarker-guided strategy based on specific non-invasive biomarkers as defined in EUTRAIN-1 study on the basis of its detection and prediction capacities for rejection at M3 to decide whether a biopsy is performed. At M12 a routine biopsy is performed.
  Visits with biopsies for clinical indication are left to the appreciation of the investigator
  Interventions: Biological: biomarker-guided strategy

INTERVENTIONS:
Biological: biomarker-guided strategy — Patients will follow a biomarker-guided strategy based on specific non-invasive biomarkers as defined in EUTRAIN-1 study on the basis of its detection and prediction capacities for rejection at M3 to decide whether a biopsy is performed. At M12 a routine biopsy is performed
  Arms: biomarker guided follow-up

SUMMARY:
The investigator hypothesize that the combined use of (1) non-invasive biomarkers in peripheral blood predicting anti-donor immunological activation or quiescence (2) interactive and actionable data analytics delivered at the bedside will promote safe clinical follow-up of kidney transplant patients with less need for invasive and induced risk surveillance by allograft protocol biopsies to assess allograft rejection in clinically stable kidney transplant patients. It is therefore proposed an European, multicenter, prospective randomized comparing two strategies of follow-up: in the first, biopsies are guided by biomarkers, in the second one, a routine biopsy is performed at M3. In both groups, a biopsy is performed at M12 and whenever considered necessary by the clinician.

DETAILED DESCRIPTION:
The main objective of this study is to demonstrate the ability of use of non-invasive biomarkers to decrease the number of allograft biopsies during the first year after transplantation. 300 new transplanted patients in the 7 clinical transplant sites will be included in the prospective multicentre EU-TRAIN Impact study with centralized storage of samples in CHUN (blood mRNA), ICS (blood cellular assays), Saint -Louis Hospital (blood anti-HLA DSA, and non-HLA antibodies), INSERM (Biopsy mRNA). Recruitment of patients will start on the day of transplantation (d-8 for transplantation from living donors) and data/samples collected over the first year following transplantation. Realization of all the acts for the research are representing the usual medical practice (Standard Of Care: SOC) except six additional blood samples that will be collected and analyzed specifically for the research and additional analysis done specifically for the research on half of one of the two biopsy cores from the recipient. 3 additional blood samples from the living donor will also be collected and analyzed specifically for the research (timepoint of the sampling: anytime from 8 days to the day of transplant.

ELIGIBILITY:
Inclusion Criteria:

1. All men and women, age ≥18 years old.
2. Subject must be a recipient of a single renal transplant from a deceased or living donor.
3. Subject is willing and able to provide signed written informed consent and willing to comply with study procedures
4. Women of Childbearing Potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL]. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of clinical trial

Exclusion Criteria:

1. Subject with Hepatitis B chronic infection and/or active infection by Hepatitis C virus (positive blood PCR result at the moment of transplant).
2. Subjects with known human immunodeficiency virus (HIV) infection.
3. Patients with active systemic infection that requires the continued use of antibiotics.
4. Patients with neoplasia except localized skin cancer receiving appropriate treatment.
5. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period, women who are pregnant or breastfeeding or women with a positive pregnancy test on enrolment.
6. Subjects who are legally detained in an official institution.
7. Primary non-function or early graft loss due to mechanical/surgical complications.
8. Death within the first 6 months after transplantation.
9. Any condition that, in the opinion of the investigator, might interfere with the patient's participation in the study, poses an added risk for the patient, or confounds the assessment of the patient
10. History of multi-organ transplant (interference with rejection natural history).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
The rate of biopsies | up to 12 months
  comparison of the rate of biopsies performed during the first year in the Group of biomarkers guided biopsies vs. routine Group

SECONDARY OUTCOMES:
Rate of immunosuppressant treatment modifications | 12month
  Rate of immunosuppressant treatment modifications in both groups.
Rate of complications due to performed biopsies | 12month
  Rate of complications due to performed biopsies between both groups
Type of biopsy-proven rejections between both groups | 12month
  Type of biopsy-proven rejections between both groups at 12 months after transplantation
Severity of biopsy-proven rejections between both groups | 12month
  Severity of biopsy-proven rejections between both groups at 12 months after transplantation
Outcome of biopsy-proven rejections between both groups | 12month
  Outcome of biopsy-proven rejections between both groups at 12 months after transplantation
Incidence of death | 12 months
  Incidence of death at 12 months after transplantation
Incidence of allograft loss | 12 months
  Incidence of allograft loss at 12 months after transplantation
Economic impact of implementing biomarkers in European Healthcare systems (cost/benefit) | up to 12 months
  Economic impact of implementing biomarkers in European Healthcare systems (cost/benefit) at 12 months after transplantation
Health-related Quality of life (QoL) of transplant patients after receiving a user-friendly reporting format from the EU-TRAIN report. | 12 months
  Health-related Quality of life (QoL) of transplant patients after receiving a user-friendly reporting format from the EU-TRAIN report.

OTHER OUTCOMES:
Safety endpoint | up to 12 months
  Comparison of The mean eGFR in both Groups estimated by glomerular filtration rate (CKD-EPI eGFR) at 12 months' post-transplantation and of the number of allograft rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Pr, Study Director — APHP
Locations (8):
- France (3):
  - Nantes Hospital, Nantes
  - Saint-Louis Hospital, Paris, Paris, Île-de-France Region
  - Necker Hospital, Paris, Paris, Île-de-France Region
- Germany (2):
  - Charité-Universitätsmedizin, Berlin, Berlin
  - Charité-Universitätsmedizin,, Berlin
- Spain (2):
  - Vall d'Hebron Hospital, Barcelona
  - Bellvitge University Hospital, Barcelona
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland